CLINICAL TRIAL: NCT06388005
Title: The Application of Emotion Release Technology in Anxiety Patients Before Daytime
Brief Title: The Application of Emotion Release Technology in Anxiety Patients Before Daytime Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-060
Record Dates: First submitted 2024-04-09; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Day Surgery; Preoperative Nursing Care; Emotional Freedom Technique
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- experimental group (Experimental)
  Interventions: Other: emotional freedom technique (EFT)

INTERVENTIONS:
Other: emotional freedom technique (EFT) — The emotional freedom technique (EFT), founded by American scholar Gary Craig, is based on the methods of meridian science in traditional Chinese medicine (TCM) and Western psychology. Guided by the TCM theory of meridians, it quickly releases negative emotions by combining acupoint stimulation with neuro-linguistic programming, and its effectiveness has been confirmed by multiple studies.
  Arms: experimental group

SUMMARY:
Research methods

1 Data collection and evaluation tools

1. The general data record sheet was self-designed by the research team, and the collected content included age, gender, BMI, occupation, general family status, economic situation, history of hypertension and cardiovascular diseases, history of anxiety and depression, self-rating anxiety scale (SAS) score, blood pressure and heart rate before and after intervention, disease diagnosis and severity, etc.
2. The anxiety was self-scored using the VAS-A (0-10 points), with 0 point as no anxiety and 10 as severe anxiety.
3. Negative emotional intensity was scored using the subjective unit of disturbance scale (SUDS, 0-10 points), with 0 point as no and 10 points as severe.
4. Nursing satisfaction was scored by the self-designed questionnaire (1-5 points): 5 points, very satisfied; 4 points, relatively satisfied; 3 points, satisfied; 2 points, medium; 1 point, dissatisfied.

2 Intervention method of the control group The control group was given routine nursing. After entering the pre-anesthesia room, the patients were scored using the VAS-A, and those with VAS-A score ≥ 5 were considered to meet the inclusion criteria. After identity authentication, the preoperative precautions and reasons for waiting in the pre-anesthesia room were explained to the patients, and answers were provided to the questions raised by the patients. After routine nursing, VAS-A score was recorded, blood pressure and heart rate were monitored, and nursing satisfaction was inquired. The survey of patient satisfaction with nursing was completed before entering the operating room.

3 Intervention method of the experimental group 3.1 Researcher training Before intervention, 4 nurses were trained for 5 d by a nurse with EFT qualification certificate, 1 h per day. The training content included: theoretical knowledge of EFT, tapping techniques, etc. After training, two assessments were conducted. Only those who scored above 90 points in both assessments could participate in the study.

3.2 Operating instructions The acupoint diagram was distributed to the experimental group by nurses, and the essentials and precautions of acupoint tapping were explained. The nurses demonstrated and tapped the acupoints on the patients while explaining, and then instructed them to tap on their own until they were able to complete the task independently and proficiently. For patients with upper limb vein puncture, proper fixation and close observation were needed, and the flexible nature of the puncture needle that would not affect operations was explained to the patients to eliminate their concerns.

3.3 Intervention content After routine nursing, the patients received EFT intervention. In addition, subjective anxiety was scored, blood pressure and heart rate were monitored, and nursing satisfaction was surveyed after admission and intervention. The specific methods are as follows.

1. Preparation stage The patients with VAS-A score ≥ 5 meeting the inclusion criteria were in a comfortable position with eyes closed, and adopted breathing exercise to relax their whole body. The patients were guided to summarize the main current distresses, such as fear, tension, pain, surgical prognosis, economic burden, etc., name the caused negative emotions, and use the SUDS to evaluate the intensity of negative emotions. The patients were asked to recite silently the prompt "Although I am very ** (a negative emotional word) now, I still deeply and completely love and accept myself" while tapping.
2. Tapping stage The patients were guided to gently massage the sore points on both sides of the body (2-3 fingers below the midpoint of the clavicle) with their five fingers together in a clockwise direction, while silently reciting the prompt 3 times. Then, the patients were guided to close their index and middle fingers together and gently tap the Zanzhu, Tongziliao, Chengqi, Renzhong, Chengjiang, Shufu, Dabao and Baihui acupoints successively with their fingertips at 2-3 times/s and the force they can bear. The prompt was recited silently when tapping each acupoint. After 3-5 rounds of tapping, 3 deep breaths were taken to re-evaluate the intensity of negative emotions.
3. Feedback stage After tapping, the patients communicated with the nurses at least once about their evaluated negative emotional intensity score and whether the score was accepted. If the tapping effect was not obvious, the evaluation was conducted by nurses, and the patients were guided to massage the sore points while silently reciting the prompt 3 times. To relieve reverse psychological drive, tapping was continued until the intensity of negative emotions reduced.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-64 years;
* preoperative visual analog scale-anxiety (VAS-A) score (0-10 points) ≥ 5 points;
* patients volunteer to participate in this study and signing the informed consent.

Exclusion Criteria:

* mental disorders, disorders of consciousness;
* restricted movement of the upper limbs and hands;
* history of hypertension;
* severe complications of the heart, brain and kidney;
* history of anxiety, long-term use of anti-anxiety and anti-depression drugs.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
VAS-A score | before and 5 min after intervention
  The anxiety was self-scored using the VAS-A (0-10 points), with 0 point as no anxiety and 10 as severe anxiety.
hemodynamic and endocrine indicators | before and 5 min after intervention
  Hemodynamic and endocrine indicators includes systolic blood pressure, diastolic blood pressure, and heart rate
nursing satisfaction | After nursing
  Nursing satisfaction was scored by the self-designed questionnaire (1-5 points): 5 points, very satisfied; 4 points, relatively satisfied; 3 points, satisfied; 2 points, medium; 1 point, dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China